CLINICAL TRIAL: NCT04892901
Title: Effectiveness of Erector Spinae Plane Block in Uniportal VATS Lung Resections
Brief Title: Erector Spinae Plane Block in Uniportal VATS
Acronym: ESPB-UVATS
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3921
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2023-12

CONDITIONS: Thoracic Surgery; Uniportal Video Assisted Thoracic Surgery (U-VATS); Lung Resections; Post-Operative Pain, Chronic; Acute Pain; Post-operative Complications; Locoregional Anesthesia
Keywords: ESPB; Erectus Spinae Plane Block; SAPB; Serratus Anterior Plane Block; ICNB; Intercostal Block; Uniportal VATS; Thoracic Surgery
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- c-ESPB group: Postoperative analgesia ensured by continuous ultrasound-guided ESPB performed at the end of surgery.
  Interventions: Procedure: c-ESPB
- c-SAPB group: Postoperative analgesia ensured by continuous SAPB performed by surgeons at the end of surgery.
  Interventions: Procedure: c-SAPB
- ICNB-group: Postoperative analgesia ensured by "one-shot" ICNB + continuous intravenous administration of tramadol by elastomeric pump.
  Interventions: Procedure: ICNB

INTERVENTIONS:
Procedure: c-ESPB — In the c-ESPB group an ultrasound-guided ESPB will be performed by the attending anaesthesiologist at the end of surgery, immediately after the last surgical stitch and before extubation. After an initial bolus of 20 ml 0,2% ropivacaine, a catheter will be left in place into the fascial plane deep to the erector spinae muscle to ensure continuous infusion (5ml/h for 48 hours) of the local anesthetic.
  Groups: c-ESPB group
Procedure: c-SAPB — In the c-SAPB group SAPB will be performed by surgeons intraoperatively, immediately before the closure of chest wall muscle planes, by injection of 20 ml 0,2% ropivacaine into the fascial plane above the Serratus Anterior muscle. After the initial bolus, a catheter will be left in place into the superficial fascial plane of the Serratus Anterior muscle to ensure continuous infusion (5ml/h for 48 hours) of the local anesthetic.
  Groups: c-SAPB group
Procedure: ICNB — In the ICNB-group ICNB will be performed by surgeons intraoperatively, immediately before chest drain placement, by injection of 20 ml of 0,2% ropivacaine into the intercostal spaces (III-VII), below the parietal pleura, under direct visualization of the neurovascular bundle. The "one-shot" ICNB will be associated in this group with intravenous administration of tramadol (300 mg/48 h) by elastomeric pump.
  Groups: ICNB-group

SUMMARY:
The main aim of this study is to compare the effectiveness of three alternative techniques (continuous Erectus Spinae Plane Block : c-ESPB; continuous Serratus Anterior Plane Block : c-SAPB; and Intercostal Nerve Block: ICNB) in reducing the severity of early postoperative pain after Uniportal-VATS lung resections. Primary outcomes will be opioid and other analgesic drugs consumption in the 72 hours after surgery, and static and dynamic pain scores, measured by the visual analog scale (VAS), at 6 pre-established time-points during the first 48 hours postoperatively. Further outcomes will be incidence of pulmonary and cardiac complications until patient's discharging, pain when removing drains, presence/absence of chronic neuropathic pain (12 weeks after surgery).

DETAILED DESCRIPTION:
Patients will be enrolled into three groups:

1. continuous Erector Spinae Plane Block group (c-ESPB group)
2. continuous Serratus Anterior Plane Block group (c-SAPB group)
3. Intercostal Nerve Block group (ICNB group)

   * In the c-ESPB group an ultrasound-guided ESPB will be performed by the attending anaesthesiologist at the end of surgery, immediately after the last surgical stitch and before extubation. After an initial bolus of 20 ml 0,2% ropivacaine, a catheter will be left into the fascial plane deep to the erector spinae muscle to ensure continuous infusion (5ml/h for 48 hours) of the local anesthetic.
   * In the c-SAPB group SAPB will be performed by surgeons intraoperatively, immediately after chest wall disclosure, by injection of 20 ml 0,2% ropivacaine into the fascial plane deep to the Serratus Anterior muscle. After the initial bolus, a catheter will be left into the fascial plane deep to the Serratus Anterior muscle to ensure continuous infusion (5ml/h for 48 hours) of the local anesthetic.
   * In the ICNB-group ICNB will be performed by surgeons intraoperatively, immediately after drain placement, by injection of 20 ml of 0,2% ropivacaine from within the chest under direct visualization of the intercostal spaces. The "one-shot" ICNB will be associated in this group with intravenous administration of tramadol (300 mg/48 h) by elastomeric pump.

The enrollment of patients into a specific group will depend on surgical variables (like disruption or not of serratus muscle/intercostal fascial planes), availability of an operator (surgeon/anesthesiologist) skilled in performing peripheral nerve blocks, logistic variables (availability of materials and ultrasound equipment).

The above mentioned primary/secondary outcome measures will be evaluated in each group and compared among them.

ELIGIBILITY:
Inclusion Criteria:

• Age >18 years

Exclusion Criteria:

* Patients who will not sign the informed consent.
* Patients scheduled for open thoracic surgery or not undergoing Uniportal-VATS resections.
* Patients undergoing concomitant chest wall, diaphragm resection or mechanical/chemical pleurodesis.
* History of previous thoracic surgery.
* Patients with Chronic Post-Thoracotomy Pain.
* Rib cage deformity or scoliosis.
* Inherited or acquired coagulopathies.
* History of allergy to drugs used during the study.
* Age < 18 years.
* Patients suffering from psychiatric or neurodegenerative diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients (age > 18 years) scheduled for Uniportal-VATS lung resections, regardless of whether for benign or malignant disease and for any type of lung resection (segmentectomy, lobectomy, atypical lung resection).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
analgesic drug consumption | first 72 hours after extubation
  number of doses of analgesic drugs administered on patients' request during the postoperative period
severity of early postoperative pain | first 48 hours after extubation
  static and dynamic pain scores, measured by the visual analog scale (VAS), at 6 pre-established time-points during the first 48 hours postoperatively.

SECONDARY OUTCOMES:
respiratory and cardiac complications | first 72 hours after extubation
  Incidence of post-operative respiratory complications (i.e. atelectasis, pneumonia, arrhythmias, etc)
pain at drain removal | chest drain removal (third/fourth postoperative day)
  severity of pain, measured by the visual analog scale (VAS), at chest drain removal
incidence of chronic pain | 12 weeks after surgery
  presence of chronic neuropathic pain after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dania Nachira, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS; Giovanni Punzo, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No